CLINICAL TRIAL: NCT00410046
Title: An Open-label, Multicentre, Supplementary Extension Study of Etanercept in Subjects With Ankylosing Spondylitis
Brief Title: Extension Study Evaluating Etanercept in Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881A3-405
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-04

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

ARMS (1):
- Etanercept (ETN) (Experimental): Patients received ETN dose 50 mg once weekly or Sulphasalazine dose 3 g daily in study 402 for 16 weeks. Upon enrollment into study 405, all received subcutaneous injections of etanercept 50 mg once weekly for 36 weeks.
  Interventions: Drug: Enbrel (etanercept)

INTERVENTIONS:
Drug: Enbrel (etanercept) — Etanercept 50 mg SC injection once weekly
  Other Names: Enbrel

SUMMARY:
The primary purpose of this study is to evaluate the health care resource utilization and work status of patients with ankylosing spondylitis undergoing treatment with etanercept by comparing study evaluations with the baseline evaluations in the ASCEND (0881A3-402)(NCT00247962) study.

ELIGIBILITY:
Inclusion criteria:

* Patients who completed 16 weeks of treatment and have completed the baseline health care resource utilization questionnaire at screening in the ASCEND study 0881A3-402-WW from participating countries.

Exclusion criteria:

* Withdrawal from the ASCEND study for safety or any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth Reserach
Locations (16):
- Denmark (4):
  - Fredriksberg
  - Odense
  - Svendborg
  - Vejle
- Finland (4):
  - Helsinki
  - Hyvinkää
  - Kuopio
  - Tampere
- Stockholm, Sweden
- United Kingdom (7):
  - Basingstoke
  - Bath
  - Cambridge
  - Cannock
  - Liverpool
  - Metropolitan Borough of Wirral
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Baraliakos X, Szumski AE, Kwok KK, Vlahos B, Borlenghi CE. Long-term Etanercept Response for Patients with Radiographic Axial Spondyloarthritis Based on Achievement of Early, Intermediate, or Late Responses During Index Studies. Rheumatol Ther. 2024 Jun;11(3):583-597. doi: 10.1007/s40744-024-00656-3. Epub 2024 Mar 15. PMID 38488976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Europe from November 2006 to January 2008.
Pre-assignment Details: Patients in 0881A3-402 (NCT00247962) were randomized to receive etanercept (ETN) or sulphasalazine (SSZ). After completion, they were eligible for enrollment into this extension study and all patients received ETN. Outcome measure analysis kept the 0881A3-402 assignment of ETN or SSZ. This enabled an analysis of changes from the original baseline.
Groups:
- Etanercept: Patients received ETN dose 50 mg once weekly or Sulphasalazine dose 3 g daily in study 0881A3-402 for 16 weeks. Upon enrollment into this study, all received subcutaneous injections of etanercept 50 mg once weekly for 36 weeks.
Period: Overall Study
Arm/Group | Etanercept
Started | 84
Completed | 79
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 42.70 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 71

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients Utilizing Healthcare Resources During 48 Weeks of Treatment
Description: Healthcare resources were defined as hospital admissions, therapeutic warm baths, physiotherapist visits, and outpatient physician visits. Healthcare resource utilization was evaluated using a questionnaire asking patients whether or not they had used the healthcare resource during the 48 weeks of treatment.
Time Frame: 48 weeks
Population: All patients who completed study 0881A3-402 (NCT00247962), continued into this study, received at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Number; unit: patients
Groups:
- Etanercept / ETN: Patients received ETN dose 50 mg once weekly in study 0881A3-402 for 16 weeks. Upon enrollment into study 405, all received subcutaneous injections of etanercept 50 mg once weekly for 36 weeks.
- SSZ / ETN: Patients received Sulphasalazine dose 3 g daily in study 0881A3-402 for 16 weeks. Upon enrollment into study 405, all received subcutaneous injections of etanercept 50 mg once weekly for 36 weeks.
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 59 | 25
patients
  Admissions to hospital | 4 | 2
  Therapeutic warm bath sessions | 4 | 4
  Physiotherapist visits | 11 | 6
  Out-patient physician visit | 30 | 10
Statistical Analysis 1: Comparison: Etanercept / ETN vs SSZ / ETN; Admissions to hospital; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept / ETN vs SSZ / ETN; Therapeutic warm bath sessions; Test type: Superiority or Other; p = 0.23, Fisher Exact
Statistical Analysis 3: Comparison: Etanercept / ETN vs SSZ / ETN; Physiotherapist visits; Test type: Superiority or Other; p = 0.567, Fisher Exact
Statistical Analysis 4: Comparison: Etanercept / ETN vs SSZ / ETN; Out-patient physician visit; Test type: Superiority or Other; p = 0.475, Fisher Exact

2. Secondary Outcome: Number of Times Healthcare Resources Were Used Per Patient During 48 Weeks of Treatment
Description: Healthcare resources were defined as hospital admissions, therapeutic warm baths, physiotherapist visits, and outpatient physician visits. Healthcare resource utilization was evaluated using a questionnaire asking all patients whether or not they had used the healthcare resource during the 48 weeks of treatment, and if so, how many times the resource was used. The mean number of times is based on those patients who responded to the questionnaire stating they had utilized healthcare resources (see outcome measure 3).
Time Frame: 48 weeks
Population: All patients who completed study 0881A3-402 (NCT00247962), continued into study 0881A3-405, received at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Mean (Full Range); unit: # of times utilized per patient
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 59 | 25
# of times utilized per patient
  Inpatient hospitalization days per patient | 6.13 [0.50 to 12.00] | 2.75 [0.50 to 5.00]
  Therapeutic warm bath sessions per patient | 6.13 [0.50 to 15.00] | 14.00 [5.00 to 26.00]
  Physiotherapist visits per patient | 11.41 [0.50 to 30.00] | 16.58 [0.50 to 43.00]
  Out-patient physician visit per patient | 2.08 [0.50 to 10.00] | 2.4 [0.00 to 6.00]
Statistical Analysis 1: Comparison: Etanercept / ETN vs SSZ / ETN; Inpatient hospitalization days per patient; Test type: Superiority or Other; p = 0.628, ANCOVA; One-way ANCOVA, baseline was a covariate
Statistical Analysis 2: Comparison: Etanercept / ETN vs SSZ / ETN; Therapeutic warm bath sessions per patient; Test type: Superiority or Other; p = 0.045, ANCOVA
Statistical Analysis 3: Comparison: Etanercept / ETN vs SSZ / ETN; Physiotherapist visits per patient; Test type: Superiority or Other; p = 0.361, ANCOVA
Statistical Analysis 4: Comparison: Etanercept / ETN vs SSZ / ETN; Out-patient physician visit per patient; Test type: Superiority or Other; p = 0.816, ANCOVA

3. Secondary Outcome: Number of Patients With Sick Leave During 48 Weeks Treatment
Description: The impact of treatment on work productivity was assessed by sick leave. Patients were asked whether or not they had taken sick leave during the 48 weeks of treatment, and if so, how many days.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 59 | 25
patients
  Patients employed during the study | 45 | 13
  Patients with sick leave during the past 12 months | 23 | 10
Statistical Analysis 1: Comparison: Etanercept / ETN vs SSZ / ETN; Analysis completed for patients with sick leave during the past 12 months; Test type: Superiority or Other; p = 1.00, Fisher Exact

4. Secondary Outcome: Number of Sick Days Per Patient During the 48 Weeks of Treatment
Description: Patients were asked whether or not they had taken sick leave during the 48 weeks of treatment, and if so, how many days. The mean number of days is based on those patients who had sick leave during the treatment period.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: Sick days per patient
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 59 | 25
Sick days per patient | 37.67 [0.50 to 232.00] | 40.05 [2.00 to 252.00]
Statistical Analysis 1: Comparison: Etanercept / ETN vs SSZ / ETN; Test type: Superiority or Other; p = 0.906, ANCOVA

5. Secondary Outcome: Change in Patient Global Assessment of Disease Activity From Baseline to Week 38
Description: Patient Global Assessment of Disease Activity was measured on a 0 to 100 mm Visual Analog Scale (VAS), with 0 mm = no disease activity. The 0881A3-402 (NCT00247962) baseline score was used as the baseline for this analysis. Change = baseline - week 38.
Time Frame: Baseline and 38 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 52 | 24
units on scale | 46.23 (24.24) | 36.08 (36.09)

6. Secondary Outcome: Change in Total Back Pain Score From Baseline to Week 38
Description: Total Back Pain was measured on a 0 to 100 mm VAS, with 0 mm indicating no pain. The 0881A3-402 (NCT00247962) baseline score was used as the baseline for this analysis. Change = baseline - week 38.
Time Frame: Baseline and 38 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 52 | 24
units on scale | 41.06 (28.52) | 34.17 (31.40)

7. Secondary Outcome: Change in Bath Ankylosing Spondylitis Functional Index (BASFI) Score From Baseline to Week 38
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in Ankylosing Spodylitis (AS) patients. Utilizing a VAS of 0-10 (0=easy, 10=impossible), patients answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a mean score of the 10 questions, with a maximum score of 100 mm. The 0881A3-402 (NCT00247962) baseline score was used as the baseline for this analysis. Change = baseline - week 38.
Time Frame: Baseline and 38 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 52 | 24
units on scale | 32.95 (20.81) | 23.41 (21.14)

8. Secondary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score From Baseline to Week 38
Description: BASDAI is a validated self assessment tool used to determine disease activity in patients with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) patient's answered 6 questions measuring discomfort, pain and fatigue. The final BASDAI score averages the individual assessments for a final score range of 0-10. The 0881A3-402 (NCT00247962) baseline score was used as the baseline for this analysis. Change = baseline - week 38.
Time Frame: Baseline and 38 weeks
Population: All patients who received at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 52 | 24
units on scale | 46.00 (31.45) | 31.13 (43.76)

9. Primary Outcome: Number of Patients Using Healthcare Resources in the 48 Weeks Before and During Treatment
Description: Healthcare resources were defined as hospital admissions, therapeutic warm baths, physiotherapist visits, and outpatient physician visits. Healthcare resource utilization was evaluated using a questionnaire asking patients whether or not they had used the healthcare resource during the 48 weeks preceding enrollment in study 0881A3-402 (NCT00247962) and during the 48 weeks of treatment in this extension study (0881A3-405).
Time Frame: 96 weeks
Population: All patients who took ETN and completed study 0881A3-402 (NCT00247962), continued into this study, received at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Number; unit: patients
Arm/Group | Etanercept / ETN
Number analyzed (Participants) | 59
patients
  Hospitalization 48 weeks before treatment | 6
  Hospitalization during 48 treatment weeks | 4
  Therapeutic warm bath 48 weeks before treatment | 8
  Therapeutic warm bath during 48 treatment weeks | 4
  Visit to physiotherapist 48 weeks before treatment | 26
  Visit to physiotherapist during 48 treatment weeks | 11
  Out-patient physician 48 weeks before treatment | 40
  Out-patient physician during 48 treatment weeks | 30
Statistical Analysis 1: Comparison: Etanercept / ETN; Test type: Superiority or Other; p = 0.743, Fisher Exact — Comparison of Hospitalization 48 weeks before treatment Vs. Hospitalization during 48 treatment weeks
Statistical Analysis 2: Comparison: Etanercept / ETN; Comparison of percentages; Test type: Superiority or Other; p = 0.362, Fisher Exact — Comparison of Therapeutic warm bath 48 weeks before treatment Vs. Therapeutic warm bath during 48 treatment weeks
Statistical Analysis 3: Comparison: Etanercept / ETN; Test type: Superiority or Other; p = 0.005, Fisher Exact — Comparison of Visit to physiotherapist 48 weeks before treatment Vs. Visit to physiotherapist during 48 treatment weeks
Statistical Analysis 4: Comparison: Etanercept / ETN; Test type: Superiority or Other; p = 0.091, Fisher Exact — Comparison of Out-patient physician 48 weeks before treatment Vs. Out-patient physician during 48 treatment weeks

10. Primary Outcome: Number of Patients Taking Sick Leave in the 48 Weeks Before and During Treatment
Description: Patients were asked whether or not they had taken sick leave during the 48 weeks preceding enrollment in study 0881A3-402 (NCT00247962) and during the 48 weeks of treatment in this extension study (0881A3-405).
Time Frame: 96 weeks
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Etanercept / ETN
Number analyzed (Participants) | 59
patients
  Sick leave 48 weeks before treatment | 27
  Sick leave during 48 weeks of treatment | 23
Statistical Analysis 1: Comparison: Etanercept / ETN; Test type: Superiority or Other; p = 0.576, Fisher Exact — Comparison of Sick leave 48 weeks before treatment Vs. Sick leave during 48 weeks of treatment

11. Secondary Outcome: Change in Bath Ankylosing Spondylitis Metrology Index (BASMI) Score From Baseline to Weeks 38
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10. The 0881A3-402 (NCT00247962) baseline score was used as the baseline for this analysis. Change = baseline - week 38.
Time Frame: Baseline and 38 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 57 | 24
units on scale | 1.21 (1.40) | 0.83 (1.31)

12. Secondary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score for Fatigue From Baseline to Week 38
Description: BASDAI is a validated self assessment tool used to determine disease activity in patients with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) patient's answered 6 questions measuring discomfort, pain and fatigue. The fatigue-specific score is presented here. The 0881A3-402 (NCT00247962) baseline score was used as the baseline for this analysis. Change = baseline - week 38.
Time Frame: Baseline and 38 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 52 | 24
units on scale | 40.46 (25.53) | 29.88 (34.33)

13. Secondary Outcome: Change in Baseline Ankylosing Spondylitis Quality of Life (ASQoL) Score From Baseline to Week 38
Description: ASQoL is a questionnaire that assesses disease-specific quality of life (QoL). It consists of 18 statements that are relevant to the physical and mental conditions for a patient with Ankylosing Spondylitis (AS): mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each statement is answered by the patient as a 'Yes' (scored as 1) or 'No' (scored as 0). All item scores are summed to give a total score. Total score can range from 0 (good QoL) to 18 (poor QoL). The 0881A3-402 baseline score was used as the baseline for this analysis. Change = baseline - week 38.
Time Frame: Baseline and 38 weeks
Population: All patients who completed study 0881A3-402 (NCT00247962), continued into this study, received at least 1 dose of study drug, had at least 1 post-baseline assessment, and completed 38 weeks.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 28 | 15
units on scale | 7.64 (5.88) | 4.40 (6.19)

14. Secondary Outcome: Change From Baseline Haywood Quality of Life Score From Baseline to Week 38
Description: Haywood quality of life instrument was utilized in the United Kingdom as the ASQoL measure. The ASQoL is an AS-specific measure of QoL, scores range from 0 (good QoL) to 80 (poor QoL). ASQoL is intended to measure the quality of life by means of questions about mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Patient's 0881A3-402 baseline score was used in the analysis. Change=baseline-week 38.
Time Frame: Baseline and 38 weeks
Population: All patients from United Kingdom sites who completed study 0881A3-402 (NCT00247962), continued into this study, received at least 1 dose of study drug had at least 1 post-baseline assessment and completed 38 weeks.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept / ETN | SSZ / ETN
Number analyzed (Participants) | 27 | 14
units on scale | 25.98 (16.51) | 16.14 (19.25)

ADVERSE EVENTS:
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 5/84
Other Adverse Events (participants affected / at risk) | 66/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=84)
Liver function test abnormal (Hepatobiliary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ileitis (Gastrointestinal disorders) | 1
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=84)
Accidental injury (General disorders) | 6
Flu syndrom (General disorders) | 5
Headache (General disorders) | 6
Infection (General disorders) | 10
Injection site reaction (General disorders) | 5
Pain (General disorders) | 5
Digestive system general (Gastrointestinal disorders) | 12
Hemic and lymphatic system general (Blood and lymphatic system disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 7
Nervous system general (Nervous system disorders) | 8
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6
Upper respiratory system general (Respiratory, thoracic and mediastinal disorders) | 23
Skin and appendages general (Skin and subcutaneous tissue disorders) | 6
Iritis (Eye disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.